CLINICAL TRIAL: NCT03904056
Title: ETDRS Panretinal Photocoagulation (PRP) Combined With Intravitreal Ranibizumab (IVR) Versus Retinal Photocoagulation Targeted to Ischemic Retina Combined With IVR for the Treatment of Proliferative Diabetic Retinopathy
Brief Title: ETDRS PRP With IVR Versus Retinal Photocoagulation Targeted to Ischemic Retina With IVR for the Treatment of PDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: São Paulo State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4160/2014
Record Dates: First submitted 2019-02-11; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic Retinopathy; Macular Edema
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ETDRS-PRP group (Active Comparator): Patients with proliferative diabetic retinopathy submitted to panretinal photocoagulation (PRP) as described in ETDRS Study combined with intravitreal injection of ranibizumab (IVR) (ETDRS-PRP group) if angluofluoresceinography demonstrated the presence of actively leaking retinal neovascularization or SD-OCT demonstrated a CSFT of more than 300 µm.
  Interventions: Procedure: ETDRS-PRP group
- ISQ-RP group (Experimental): Patients with proliferative diabetic retinopathy submitted to retinal photocoagulation targeted to ischemic retina combined with intravitreal injection of ranibizumab (IVR) if angluofluoresceinography demonstrated the presence of actively leaking retinal neovascularization or SD-OCT demonstrated a CSFT of more than 300 µm.
  Interventions: Procedure: ISQ-RP

INTERVENTIONS:
Procedure: ISQ-RP — Patients were treated with single-spot targeted retinal photocoagulation directed toward areas of retinal nonperfusion detected by fluorescein angiography. In this group, laser treatment was performed in two sessions (week 0 and 2), with a shot duration of 100 ms, but spots were placed 1/2 burn apart and power modulated in order to generate moderately white spots on the retina.
  Retinal photocoagulation was performed with single-spot full-scatter PRP using Purepoint green diode laser (Alcon, Fortworth, Texas) with an Ocular Mainster PRP 165 lens with a dynamic field of view of 180 degrees, and a 200 micron spot size (which produces a 392 micron spot size on the retina). Intravitreal injection of 0.5 mg (0.05 ml) ranibizumab (Lucentis®) (IVR) were performed 180 minutes after the first laser session (week 0) by a single retina specialist.
  Other Names: intravitreal injection of ranibizumab (IVR)
  Arms: ISQ-RP group
Procedure: ETDRS-PRP group — Panretinal photocoagulation (PRP) as described in ETDRS Study combined with intravitreal injection of ranibizumab
  Arms: ETDRS-PRP group

SUMMARY:
Purpose: To compare panretinal photocoagulation (PRP) as described in ETDRS Study combined with intravitreal injection of ranibizumab (IVR) (ETDRS-PRP group) and retinal photocoagulation targeted to ischemic retina combined with IVR (ISQ-RP group) in patients with proliferative diabetic retinopathy (PDR).

Design: Randomized prospective clinical trial. Methods: Patients with PDR were assigned to receive either PRP plus IVR (20 eyes) or retinal photocoagulation targeted to ischemic areas plus IVR (20 eyes). ETDRS best-corrected visual acuity (BCVA), central subfield macular thickness (CSFT) measured by optical coherence tomography (OCT) were performed at baseline and every 4 weeks through week 48. Area of fluorescein leakage from active new vessels (FLA) was measured every 12 weeks. Full-field electroretinography (ERG) was recorded at baseline and after 3 months.

DETAILED DESCRIPTION:
This parallel clinical trial was approved by the local Research Ethics Committee, and all subjects gave written informed consent to participate. Between August 2014 and July 2016, all adult patients with treatment-naive PDR and a best-corrected visual acuity (BCVA) better than 20/800 evaluated at our facility were invited to participate in the study.

During the recruitment phase, twenty-three consecutive patients who met the inclusion and exclusion criteria were enrolled into the study. At baseline visit, each patient underwent detailed ophthalmologic assessment including BCVA measurement according to standardized ETDRS refraction protocols using modified ETDRS cards 1, 2 and R; applanation tonometry; slit-lamp biomicroscopy examination under mydriasis (including classification of crystalline lens opacity status using the Lens Opacities Classification System - LOCS III) (13); and indirect funduscopic examination. Digital ocular stereoscopic fundus photographs (TRC-50DX - IMAGEnet; Topcon, Tokyo, Japan), wide field fluorescein angiography and spectral domain optical coherence tomography (SD-OCT) (HRA-OCT, Heidelberg, Germany) were also performed.

Randomization and treatment groups

Patients were randomly assigned using a computer-generated sequence, to one of the following two treatment groups:

ETDRS-PRP Group: patients were treated in two sessions (week 0 and week 2) of 800-900 shots, for a total of 1600-1800 shots with a shot duration of 100 ms and power modulated in order to generate moderately white spots on the retina.

ISQ-RP Group: patients were treated with single-spot targeted retinal photocoagulation directed toward areas of retinal nonperfusion detected by fluorescein angiography. In this group, laser treatment was also performed in two sessions (week 0 and 2), with a shot duration of 100 ms, but spots were placed 1/2 burn apart and power modulated in order to generate moderately white spots on the retina.

For both groups, retinal photocoagulation was performed with single-spot full-scatter PRP using Purepoint green diode laser (Alcon, Fortworth, Texas) with an Ocular Mainster PRP 165 lens with a dynamic field of view of 180 degrees, and a 200 micron spot size (which produces a 392 micron spot size on the retina). Intravitreal injection of 0.5 mg (0.05 ml) ranibizumab (Lucentis®) (IVR) were performed 180 minutes after the first laser session (week 0) by a single retina specialist.

Intravitreal injection Intravitreal injections were performed in a clinic setting 180 minutes after retinal photocoagulation with a disposable syringe with a BD Ultra-FineTM 29G ½" needle, via the pars plana 3.5 mm posterior to the limbus, using topical anesthesia. After the procedure, optic nerve perfusion was assessed by indirect binocular ophthalmoscopy, with paracenthesis of the anterior chamber considered in cases of poor perfusion. After injection, patients were instructed to use antibiotic eyedrops (0.5% moxifloxacin), according to drug label, one drop every 4 hours for one week, in the eye which received the intravitreal injection.

Ophthalmologic evaluations Comprehensive ophthalmic evaluations, including ETDRS BCVA and central subfield macular thickness (CSFT) measured by SD-OCT as described elsewhere (15) were performed at baseline and every 4 weeks through week 48.

Area of fluorescein leakage from active new vessels (FLA) was measured by wide field fluorescein angiography at baseline and at weeks 4, 8, 12, 24, 36 and 48 using fluorescein angiography pictures taken 2.0 to 3.0 minutes after the injection of fluorescein dye. Local and systemic adverse effects, including changes in intraocular pressure and in crystalline lens status, were monitored throughout the study.

Retreatment criteria At follow-up visits from week 12 to 48, patients were treated quarterly with an IVR (0.5 mg in 0.05 ml) if FA demonstrated the presence of actively leaking retinal neovascularization. From weeks 4 to 48, patients could receive monthly IVR if SD-OCT demonstrated a CSFT of more than 300 µm.

ERG protocol Full-field ERG was performed at baseline, and 12, 24 and 48 weeks after treatment (ColorDome and Espion E2 - Diagnosys LLC, Middleton, MA, USA). ERG was executed in accordance to ISCEV standard [20] using DTL as positive electrodes. Skin electrodes (Red-Dot - 3M) were placed on each temporal orbital rim to serve as references, and on forehead as ground. A- and b-wave amplitude and implicit time were evaluated.

After 30 min dark adaptation, a series of flashes with increasing luminance was used as light stimuli: 0.003, 0.01 (rod ERG), 0.03, 0.1, 0.3, 1.0, 3.0 (combined rod-cone ERG) and 10 cd.s/m2. Oscillatory potentials were filtered out of combined rod-cone ERG, using an off-line fast-Fourrier algorithm set as a band-pass frequency filter (75 - 300 Hz) as previously described [21], and area under the curve (OP-AUC) between a- and b-wave implicit time was calculated.

Thereafter, patients were light adapted for 10 min, and photopic ERG measurements were also performed a series of increasing stimuli luminance: 0.1, 0.3, 1.0, 3.0 (cone ERG), 10.0 and 30.0 cd.s/m2, followed by the 30 Hz flicker (background during photopic stimulation = 30 cd/m2).

Sample size

The sample size estimation was based on the standard deviation of fluorescein leakage area of a previous study where PRP plus ranibizumab was used for proliferative diabetic retinopathy treatment (11). Considering this previous study, with a sample size of 15 patients per group, there is an 80% power to detect a mean difference of 2 mm2 between both groups.

Statistics Baseline data were compared using one-way analysis of variance followed by Tukey-Kramer testing for multiple mean comparisons, while group comparisons during follow-up were performed using analysis of covariance (ANCOVA) with "group", "time" and "group cross time" as effects, followed by Tukey HSD testing. Calculations were performed using JMP 10.0 (SAS). The significance level was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with treatment-naive PDR and a best-corrected visual acuity (BCVA) better than 20/800

Exclusion Criteria:

* Presence of advanced PDR, i.e., vitreous hemorrhage that would prevent documentation of the fundoscopic examination or administration of PRP, or presence of traction retinal detachment;
* presence of ring-shaped retinal neovascularization extending along both temporal arcades and the optic disc;
* an abnormality of the vitreoretinal interface in the macular region that would lead the investigator to consider the necessity of pars plana vitrectomy;
* intravitreal injection of corticosteroids or other antiangiogenic drugs during the prior 6 months;
* inability of patient to fixate and perform reliable automated static perimetry;
* cataract surgery during the prior 3 months;
* history of pars plana vitrectomy or scleral buckle;
* acute ocular infection;
* allergy to fluorescein;
* medical or psychological conditions that would prevent the patient from giving written informed consent or completing the study;
* significant uncontrolled disease that, in the opinion of the investigator, would prevent the patient from completing the study;
* participation in another clinical study during the previous 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Fluorescein leakage area of active new vessels (FLA) | 48 weeks
  Compare the Area of fluorescein leakage from active new vessels in both groups in mm2 measured by wide field fluorescein angiography (Optomap 200TX; Optos PLC., Dunfermline, Scotland, United Kingdom)

SECONDARY OUTCOMES:
Best-corrected visual acuity (BCVA) | 48 weeks
  Compare the Best-corrected visual acuity (BCVA) in both groups according to standardized ETDRS refraction protocols using modified ETDRS cards
Central subfield thickness (CSFT) | 48 weeks
  Compare the Central subfield thickness (CSFT) between both groups using spectral domain optical coherence tomography (SD-OCT) (HRA-OCT, Heidelberg, Germany)
Number of Ranibizumab Intravitreal Injections | 48 weeks
  to compare the number of Ranibizumab Intravitreal Injections in both groups
Electroretinography | 48 weeks
  To compare Electroretinography response in both groups using Diagnosys LLD - Espion E2 Electroretinography System

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toscano L, Messias A, Messias K, de Cenco Lopes R, Ribeiro JAS, Scott IU, Jorge R. Proliferative diabetic retinopathy treated with intravitreal ranibizumab and photocoagulation directed at ischemic retinal areas-A randomized study. Doc Ophthalmol. 2021 Dec;143(3):313-322. doi: 10.1007/s10633-021-09848-6. Epub 2021 Aug 4. PMID 34347216